CLINICAL TRIAL: NCT03122431
Title: Relevance of Monitoring Blood Levels Compared to Salivar Levels of Drugs Used in Rheumatic Autoimmune Diseases: Adherence and Understanding the Possible Underlying Mechanisms Involved in Effectiveness and in Adverse Effects
Brief Title: Relevance of Monitoring Blood and Salivar Levels of Drugs Used in Rheumatic Autoimmune Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPLC-Rheumatic diseases
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-05

CONDITIONS: Systemic Lupus Erythematosus (SLE); Juvenile SLE; Cutaneous Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Thalidomide; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: This study includes 3 subprojects that will assess serum drug levels for efficacy and toxicity. In the first two subprojects, hydroxychloroquine will be studied in SLE population. In the third subproject, thalidomide and SLE and cutaneous lupus will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SLE/cutaneous lupus with thalidomide (Other): This subproject includes only one arm of lupus patients with active and refractory cutaneous disease and eligible for Thalidomide 100mg/day for 12 months.
  Interventions: Drug: Thalidomide
- Inactive SLE with standard dose of HCQ (Active Comparator): This subproject includes one arm of lupus patients with inactive disease, in which will be maintained on standard dose of Hydroxychloroquine (400mg/day).
  Interventions: Drug: standard dose of HCQ
- Inactive SLE with reduced dose of HCQ (Active Comparator): This subproject includes one arm of lupus patients with inactive disease: in which the dose will be reduced to 400mg 3 times a week (Hydroxychloroquine reduced).
  Interventions: Drug: Hydroxychloroquine reduced

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 100 mg/day
  Other Names: Thalidomide 100 mg
  Arms: SLE/cutaneous lupus with thalidomide
Drug: Hydroxychloroquine reduced — Hydroxychloroquine 2.5 mg/kg/day
  Other Names: HCQ reduced
  Arms: Inactive SLE with reduced dose of HCQ
Drug: standard dose of HCQ — Hydroxychloroquine 5.0 mg/kg/day
  Other Names: HCQ standard
  Arms: Inactive SLE with standard dose of HCQ

SUMMARY:
No drug treatment is completely free of risk and lack of response, adverse events and poor adherence may affect its effectiveness. Within this context, this project aims to evaluate the importance of monitoring blood levels and salivary drug used in rheumatic autoimmune diseases in the monitoring of adherence to therapy. In addition, this project intends to use the monitoring of drug levels, based on pharmacokinetic studies and pharmacokinetics/pharmacodynamics modeling, to broaden the understanding of the possible cellular, tissue and immunological mechanisms involved in efficacy and adverse effects of these drugs with the prospect of reducing the damage and maintain therapeutic efficacy. The high-performance liquid chromatography (HPLC) coupled to mass spectrometry, which will be used to evaluate hydroxychloroquine, thalidomide, glucocorticoids, is considered the gold standard technology to qualitative and quantitative analysis of drugs in blood and its comparison with the dosage in the saliva is an improvement in simplification of the process. For biological agents the focus will be on the understanding the loss of efficacy and the possible role of anti-TNF antibodies using ELISA capture methodology.This project will be divided into four sections with their respective sub-projects according to the medications that will be studied: hydroxychloroquine, thalidomide, biologic agents and glucocorticoids.

DETAILED DESCRIPTION:
No drug treatment is completely free of risk and lack of response, adverse events and poor adherence may affect its effectiveness. There is also a large inter-individual variability in response to treatments with regard to efficacy and toxicity, and for many drugs, there is also a period of weeks to months to establish its efficacy. Within this context, this project aims to evaluate the importance of monitoring blood levels and salivary drug used in rheumatic autoimmune diseases in the monitoring of adherence to therapy. In addition, this project intends to use the monitoring of drug levels, based on pharmacokinetic studies and pharmacokinetics/pharmacodynamics modeling, to broaden the understanding of the possible cellular, tissue and immunological mechanisms involved in efficacy and adverse effects of these drugs with the prospect of reducing the damage and maintain therapeutic efficacy. The high-performance liquid chromatography (HPLC) coupled to mass spectrometry, which will be used to evaluate hydroxychloroquine, thalidomide, glucocorticoids, is considered the gold standard technology to qualitative and quantitative analysis of drugs in blood and its comparison with the dosage in the saliva is an improvement in simplification of the process. The implementation of this methodology dedicated to research in our center, with the necessary training of human resources, will enable the standardization and availability of this advanced technology to other muldisciplinary projects in various areas of science. For biological agents the focus will be on the understanding the loss of efficacy and the possible role of anti-TNF antibodies using ELISA capture methodology.This thematic project will be divided into four sections with their respective sub-projects according to the medications that will be studied: hydroxychloroquine, thalidomide, biologic agents and glucocorticoids.

ELIGIBILITY:
Thalidomide subproject:

Inclusion Criteria:

* SLE diagnosis according to 1997 ACR criteria
* Active and refractory cutaneous lupus lesions
* Male gender (using contraceptive barrier method) or confirmed infertility for female gender
* Normal electroneuromyography at study entry

Exclusion Criteria:

* Alcoholism
* History of peripheral neuropathy
* Previous history of thrombophilia or positive antiphospholipid antibodies
* Renal and/or central nervous system and/or hematological activity

HCQ reduced subproject:

Inclusion Criteria:

* SLE diagnosis according to 1997 ACR criteria
* Use of hydroxychloroquine (5 to 6.5mg/kg/day) for ≥5 years
* SLEDAI-2K <4

Exclusion Criteria:

* Alcoholism
* Renal dialysis
* Concomitant infectious process
* Acute and chronic liver diseases
* Concomitant use of some drugs that interact with HCQ (cimetidine, antacids, digoxin, aminoglycosides, penicillamine, neostigmine, pyridostigmine)
* Signs of Retinopathy

HCQ high subproject:

Inclusion Criteria:

* SLE diagnosis according to 1997 ACR criteria
* No use of hydroxychloroquine for ≥ 6 months
* LES/LESJ in activity (SLEDAI≥6)

Exclusion Criteria:

* Alcoholism
* Renal dialysis
* Concomitant infectious process
* Acute and chronic liver diseases
* Concomitant use of some drugs that interact with HCQ (cimetidine, antacids, digoxin, aminoglycosides, penicillamine, neostigmine, pyridostigmine)
* Signs of Retinopathy

Ages: 5 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa Bonfa, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S, Kantor J, Kim E, Militello G, McGinnis K, Richardson S, Treat J, Vittorio C, Van Voorhees A, Werth VP. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): an outcome instrument for cutaneous lupus erythematosus. J Invest Dermatol. 2005 Nov;125(5):889-94. doi: 10.1111/j.0022-202X.2005.23889.x. PMID 16297185
- [Background] Bai N, Cui XY, Wang J, Sun CG, Mei HK, Liang BB, Cai Y, Song XJ, Gu JK, Wang R. Determination of thalidomide concentration in human plasma by liquid chromatography-tandem mass spectrometry. Exp Ther Med. 2013 Feb;5(2):626-630. doi: 10.3892/etm.2012.847. Epub 2012 Nov 30. PMID 23404219
- [Background] Bernstein HN. Ocular safety of hydroxychloroquine. Ann Ophthalmol. 1991 Aug;23(8):292-6. PMID 1952638
- [Background] Briani C, Zara G, Rondinone R, Della Libera S, Ermani M, Ruggero S, Ghirardello A, Zampieri S, Doria A. Thalidomide neurotoxicity: prospective study in patients with lupus erythematosus. Neurology. 2004 Jun 22;62(12):2288-90. doi: 10.1212/01.wnl.0000130499.91775.2c. PMID 15210897
- [Background] Coelho A, Souto MI, Cardoso CR, Salgado DR, Schmal TR, Waddington Cruz M, de Souza Papi JA. Long-term thalidomide use in refractory cutaneous lesions of lupus erythematosus: a 65 series of Brazilian patients. Lupus. 2005;14(6):434-9. doi: 10.1191/0961203305lu2124oa. PMID 16038106
- [Background] Costedoat-Chalumeau N, Amoura Z, Hulot JS, Hammoud HA, Aymard G, Cacoub P, Frances C, Wechsler B, Huong du LT, Ghillani P, Musset L, Lechat P, Piette JC. Low blood concentration of hydroxychloroquine is a marker for and predictor of disease exacerbations in patients with systemic lupus erythematosus. Arthritis Rheum. 2006 Oct;54(10):3284-90. doi: 10.1002/art.22156. PMID 17009263
- [Background] Costedoat-Chalumeau N, Pouchot J, Guettrot-Imbert G, Le Guern V, Leroux G, Marra D, Morel N, Piette JC. Adherence to treatment in systemic lupus erythematosus patients. Best Pract Res Clin Rheumatol. 2013 Jun;27(3):329-40. doi: 10.1016/j.berh.2013.07.001. PMID 24238690
- [Background] Costedoat-Chalumeau N, Dunogue B, Morel N, Le Guern V, Guettrot-Imbert G. Hydroxychloroquine: a multifaceted treatment in lupus. Presse Med. 2014 Jun;43(6 Pt 2):e167-80. doi: 10.1016/j.lpm.2014.03.007. Epub 2014 May 19. PMID 24855048
- [Background] Cuadrado MJ, Karim Y, Sanna G, Smith E, Khamashta MA, Hughes GR. Thalidomide for the treatment of resistant cutaneous lupus: efficacy and safety of different therapeutic regimens. Am J Med. 2005 Mar;118(3):246-50. doi: 10.1016/j.amjmed.2004.04.030. PMID 15745722
- [Background] Frances C, Cosnes A, Duhaut P, Zahr N, Soutou B, Ingen-Housz-Oro S, Bessis D, Chevrant-Breton J, Cordel N, Lipsker D, Costedoat-Chalumeau N. Low blood concentration of hydroxychloroquine in patients with refractory cutaneous lupus erythematosus: a French multicenter prospective study. Arch Dermatol. 2012 Apr;148(4):479-84. doi: 10.1001/archdermatol.2011.2558. PMID 22508872
- [Background] Giannini F, Volpi N, Rossi S, Passero S, Fimiani M, Cerase A. Thalidomide-induced neuropathy: a ganglionopathy? Neurology. 2003 Mar 11;60(5):877-8. doi: 10.1212/01.wnl.0000049462.03800.b1. No abstract available. PMID 12629253
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1997 Sep;40(9):1725. doi: 10.1002/art.1780400928. No abstract available. PMID 9324032
- [Background] Jallouli M, Galicier L, Zahr N, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Le Thi Huong D, Asli B, Kahn JE, Pourrat J, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Leroux G, Cohen-Bittan J, Sellam J, Mariette X, Blanchet B, Hulot JS, Amoura Z, Piette JC, Costedoat-Chalumeau N; Plaquenil Lupus Systemic Study Group. Determinants of hydroxychloroquine blood concentration variations in systemic lupus erythematosus. Arthritis Rheumatol. 2015 May;67(8):2176-84. doi: 10.1002/art.39194. PMID 25989906
- [Background] Knop J, Bonsmann G, Happle R, Ludolph A, Matz DR, Mifsud EJ, Macher E. Thalidomide in the treatment of sixty cases of chronic discoid lupus erythematosus. Br J Dermatol. 1983 Apr;108(4):461-6. doi: 10.1111/j.1365-2133.1983.tb04600.x. PMID 6838771
- [Background] Kyriakis KP, Kontochristopoulos GJ, Panteleos DN. Experience with low-dose thalidomide therapy in chronic discoid lupus erythematosus. Int J Dermatol. 2000 Mar;39(3):218-22. doi: 10.1046/j.1365-4362.2000.00953.x. PMID 10759967
- [Background] Michaelides M, Stover NB, Francis PJ, Weleber RG. Retinal toxicity associated with hydroxychloroquine and chloroquine: risk factors, screening, and progression despite cessation of therapy. Arch Ophthalmol. 2011 Jan;129(1):30-9. doi: 10.1001/archophthalmol.2010.321. PMID 21220626
- [Background] Morita S, Takahashi T, Yoshida Y, Yokota N. Population Pharmacokinetics of Hydroxychloroquine in Japanese Patients With Cutaneous or Systemic Lupus Erythematosus. Ther Drug Monit. 2016 Apr;38(2):259-67. doi: 10.1097/FTD.0000000000000261. PMID 26587870
- [Background] Tsakonas E, Joseph L, Esdaile JM, Choquette D, Senecal JL, Cividino A, Danoff D, Osterland CK, Yeadon C, Smith CD. A long-term study of hydroxychloroquine withdrawal on exacerbations in systemic lupus erythematosus. The Canadian Hydroxychloroquine Study Group. Lupus. 1998;7(2):80-5. doi: 10.1191/096120398678919778. PMID 9541091
- [Derived] Zanetti CB, Pedrosa T, Kupa LVK, Aikawa NE, Borba EF, Vendramini MBG, Silva CA, Pasoto SG, Bonfa E. Hydroxychloroquine blood levels in stable lupus nephritis under low dose (2-3 mg/kg/day): 12-month prospective randomized controlled trial. Clin Rheumatol. 2021 Jul;40(7):2745-2751. doi: 10.1007/s10067-021-05600-2. Epub 2021 Jan 24. PMID 33486596

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactive SLE With Standard Dose of HCQ: Lupus nephritis patients on stable inactive disease for at least 6 months prescribed full 2016-AAO dose of HCQ (4-5.5 mg/kg/day, real body weight).
- Inactive SLE With Reduced Dose of HCQ: Lupus nephritis patients on stable inactive disease for at least 6 months prescribed reduced 2016-AAO dose of HCQ (2-3.0 mg/kg/day, real body weight)
- SLE/Cutaneous Lupus With Thalidomide: Adult patients with CLE (biopsy proven)/SLE (American College of Rheumatology classification criteria, 1997) treated with thalidomide.
  Inclusion criteria:
  1. absence of pregnancy potential for females;
  2. agreement of male patients to use condoms throughout the treatment period with thalidomide and up to 30 days after its ending, even though they had already undergone vasectomy;
  3. active skin lesions;
  4. no response to previous use of HCQ, prednisone 20 mg/day, and immunosuppressants/dapsone or indication of thalidomide according to the attending physician; 5) agreement of recruited patients to participate in the study according to signed informed consent form, and agreement to thalidomide use according to signed responsibility term at starting treatment and at each renewal of the prescription; 6) a normal NCS;
  7) normal serum vitamin B12 levels; 8) negative tests for hepatitis B/C and HIV; 9) negative antiphospholipid antibodies.
  Exclusion criteria:
  1. other associated autoimmune diseases, such as Sjogren's syndrome;
  2. previous or current alcoholism;
  3. diabetes mellitus;
  4. history of PN;
  5. previous use of thalidomide;
  6. previous or current use of leflunomide, TNF-alpha inhibitors, chemotherapy and other neurotoxic drugs;
  7. history of cancer or thrombosis;
  8. current renal or nervous system lupus activities, autoimmune haemolytic anaemia and/or thrombocytopenia <50,000/mm3;
  9. inability to understand the study.
Period: Overall Study
Arm/Group | Inactive SLE With Standard Dose of HCQ | Inactive SLE With Reduced Dose of HCQ | SLE/Cutaneous Lupus With Thalidomide
Started | 41 | 32 | 20
Completed | 41 | 32 | 9
Not Completed | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive SLE With Standard Dose of HCQ | Inactive SLE With Reduced Dose of HCQ | SLE/Cutaneous Lupus With Thalidomide | Total
Number analyzed (Participants) | 41 | 32 | 20 | 93
Age, Continuous [Median (Standard Deviation); unit: years] | 37 (10.5) | 37 (6.9) | 44.8 (7.6) | 37 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 17 | 85
  Male | 2 | 3 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 6 | 9 | 28
  Non-Caucasian | 28 | 26 | 11 | 65
Drug blood levels [Mean (Standard Deviation); unit: ng/mL] — Population: Baseline hydroxychloroquine levels in this arm were not measured.
  ng/mL
    number analyzed (Participants) | 41 | 32 | 0 | 73
    (all) | 1343.5 (521.5) | 1404.9 (492.0) |  | 1374.2 (506.8)

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of Thalidomide
Description: Serum levels of thalidomide by liquid chromatography and tandem mass spectrometry (HPLC-MS/MS)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- SLE/Cutaneous Lupus With Thalidomide: Adult patients with CLE (biopsy proven)/SLE (American College of Rheumatology classification criteria, 1997) treated with thalidomide.
Arm/Group | SLE/Cutaneous Lupus With Thalidomide
Number analyzed (Participants) | 20
ng/mL | 415.1 (326.0)

2. Primary Outcome: Serum Levels of Hydroxycloroquine
Description: Serum levels of hydroxycloroquine by LCMS
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Inactive SLE With Standard Dose of HCQ | Inactive SLE With Reduced Dose of HCQ
Number analyzed (Participants) | 41 | 32
ng/mL | 991.6 (576.3) | 569.0 (533.4)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- SLE/Cutaneous Lupus With Thalidomide: SLE/cutaneous lupus with thalidomide arm (12 months).
Arm/Group | SLE/Cutaneous Lupus With Thalidomide | Inactive SLE With Standard Dose of HCQ | Inactive SLE With Reduced Dose of HCQ
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/41 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/41 | 0/32
Other Adverse Events (participants affected / at risk) | 12/20 | 0/41 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLE/Cutaneous Lupus With Thalidomide (N=20) | Inactive SLE With Standard Dose of HCQ (N=41) | Inactive SLE With Reduced Dose of HCQ (N=32)
Only sensory peripheral neuropathy (Nervous system disorders) | 12 (12) | 0 (0) | 0 (0) — Only sensory peripheral neuropathy evaluated by nerve conduction study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03122431/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03122431/ICF_001.pdf